CLINICAL TRIAL: NCT04203927
Title: Effects of Empagliflozin on Cardiac Microvasculature and Insulin Sensitivity in Subjects With Type 2 Diabetes
Acronym: EJB051
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Eugene Barrett, Prinicipal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 21403; 1R01HL142250-01A1 (NIH)
Record Dates: First submitted 2019-12-17; First posted 2019-12-18 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Type2 Diabetes; Insulin Sensitivity
MeSH Terms: conditions — Insulin Resistance | interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin + insulin infusion (Active Comparator): vascular measurements in overnight fasted state and during insulin infusion
  Interventions: Drug: Empagliflozin 25 MG
- Empagliflozin + mixed meal (Active Comparator): vascular measurements in overnight fasted state and 2 hours after mixed meal 10kcal/kg body weight ( 55% Cho, 30%Fat, 20% Pro)
  Interventions: Drug: Empagliflozin 25 MG

INTERVENTIONS:
Drug: Empagliflozin 25 MG — SGLT-2 inhibitor

SUMMARY:
The aim is to test in T2DM patients, whether, compared to placebo, 12 weeks of SGLT-2 inhibitor improves post-absorptive, post-insulin infusion or postprandial insulin action to enhance Cardiac Muscle vascular function and whether changes correlate with improved GV or postprandial hyperglycemia

DETAILED DESCRIPTION:
The investigators will study 32 T2DM subjects measuring cardiac muscle vascular function before and after a 4 hour insulin clamp ( protocol A) and before and after a mixed meal (protocol B). Then subjects will be randomized into 2 groups: Group 1 will undergo a 12 week intervention of Empagliflozin, and Group 2 will do 12 weeks of Placebo. The intervention will be single blinded. At the end of the 12 week intervention subjects will repeat protocol A and B.

The study's primary objective is to assess whether, compared to placebo, 12 weeks of Empagliflozin improves post-absorptive or postprandial insulin action to enhance myocardial perfusion (MP) and whether changes of MP correlate with improved glucose variability or postprandial hyperglycemia

ELIGIBILITY:
Inclusion Criteria:

* A1C > 6.5 and <9%
* Never on SGLT-2i (eg: Jardiance, Invokana, Farxiga, Steglatro)
* On stable dose of oral hypoglycemic agents >3 months
* On stable dose of other medications for >3 months
* BMI-<35

Exclusion Criteria:

* • Smoking presently or in the past 6 months

  * Taking insulin
  * BP >160/90
  * BMI >35
  * History of congestive heart failure, ischemic heart disease, severe pulmonary disease, liver or kidney disease.
  * Any vascular disease such as myocardial infarction, stroke, peripheral vascular disease
  * History of cancer or psychiatric disease
  * Presence of an intracardiac or intrapulmonary shunt (we will screen for this by auscultation during the physical exam by PI).
  * Pregnant or breastfeeding.
  * Known hypersensitivity to perflutren (contained in Definity)
  * Screening O2 saturation <90%
  * History of recurrent UTI/bladder/kidney infections-eGFR is below 45 mL/min/1.73.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Myocardial microvascular perfusion | Between baseline and 12 weeks treatment
  Vascular measure of myocardial perfusion

SECONDARY OUTCOMES:
Flow Mediated Dilation (FMD) Vascular measure of conduit artery stiffness Change in Flow Mediated Dilation (FMD) between baseline and after 2 hour insulin clamp Vascular measure of conduit artery stiffness Flow Mediated Dilation ( FMD) | Between baseline and 12 weeks of treatment.
  Vascular measure of conduit artery stiffness
Augmentation Index ( AI) | Between baseline and 12 weeks of treatment.
  Measurement of central artery stiffness
Pulse Wave Velocity ( PWV) | Between baseline and 12 weeks of treatment
  Measurement of central artery stiffness

CONTACTS AND LOCATIONS:
Overall Officials: Eugene J Barrett, MD PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Nishimura R, Tanaka Y, Koiwai K, Inoue K, Hach T, Salsali A, Lund SS, Broedl UC. Effect of empagliflozin monotherapy on postprandial glucose and 24-hour glucose variability in Japanese patients with type 2 diabetes mellitus: a randomized, double-blind, placebo-controlled, 4-week study. Cardiovasc Diabetol. 2015 Jan 30;14:11. doi: 10.1186/s12933-014-0169-9. PMID 25633683
- [Background] Inzucchi SE, Zinman B, Fitchett D, Wanner C, Ferrannini E, Schumacher M, Schmoor C, Ohneberg K, Johansen OE, George JT, Hantel S, Bluhmki E, Lachin JM. How Does Empagliflozin Reduce Cardiovascular Mortality? Insights From a Mediation Analysis of the EMPA-REG OUTCOME Trial. Diabetes Care. 2018 Feb;41(2):356-363. doi: 10.2337/dc17-1096. Epub 2017 Dec 4. PMID 29203583
- [Background] Zhao L, Chai W, Fu Z, Dong Z, Aylor KW, Barrett EJ, Cao W, Liu Z. Globular adiponectin enhances muscle insulin action via microvascular recruitment and increased insulin delivery. Circ Res. 2013 Apr 26;112(9):1263-71. doi: 10.1161/CIRCRESAHA.111.300388. Epub 2013 Mar 4. PMID 23459195
- [Background] Liu J, Jahn LA, Fowler DE, Barrett EJ, Cao W, Liu Z. Free fatty acids induce insulin resistance in both cardiac and skeletal muscle microvasculature in humans. J Clin Endocrinol Metab. 2011 Feb;96(2):438-46. doi: 10.1210/jc.2010-1174. Epub 2010 Nov 3. PMID 21047922
- [Background] Scognamiglio R, Negut C, De Kreutzenberg SV, Tiengo A, Avogaro A. Postprandial myocardial perfusion in healthy subjects and in type 2 diabetic patients. Circulation. 2005 Jul 12;112(2):179-84. doi: 10.1161/CIRCULATIONAHA.104.495127. Epub 2005 Jul 5. PMID 15998667
- [Background] Chai W, Liu J, Jahn LA, Fowler DE, Barrett EJ, Liu Z. Salsalate attenuates free fatty acid-induced microvascular and metabolic insulin resistance in humans. Diabetes Care. 2011 Jul;34(7):1634-8. doi: 10.2337/dc10-2345. Epub 2011 May 26. PMID 21617098
- [Background] Kovatchev BP, Clarke WL, Breton M, Brayman K, McCall A. Quantifying temporal glucose variability in diabetes via continuous glucose monitoring: mathematical methods and clinical application. Diabetes Technol Ther. 2005 Dec;7(6):849-62. doi: 10.1089/dia.2005.7.849. PMID 16386091
- [Background] Kovatchev BP. Metrics for glycaemic control - from HbA1c to continuous glucose monitoring. Nat Rev Endocrinol. 2017 Jul;13(7):425-436. doi: 10.1038/nrendo.2017.3. Epub 2017 Mar 17. PMID 28304392
- [Background] Zinman B, Lachin JM, Inzucchi SE. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2016 Mar 17;374(11):1094. doi: 10.1056/NEJMc1600827. No abstract available. PMID 26981940
- [Background] Neal B, Perkovic V, Matthews DR. Canagliflozin and Cardiovascular and Renal Events in Type 2 Diabetes. N Engl J Med. 2017 Nov 23;377(21):2099. doi: 10.1056/NEJMc1712572. No abstract available. PMID 29166232
- [Background] Wanner C, Inzucchi SE, Lachin JM, Fitchett D, von Eynatten M, Mattheus M, Johansen OE, Woerle HJ, Broedl UC, Zinman B; EMPA-REG OUTCOME Investigators. Empagliflozin and Progression of Kidney Disease in Type 2 Diabetes. N Engl J Med. 2016 Jul 28;375(4):323-34. doi: 10.1056/NEJMoa1515920. Epub 2016 Jun 14. PMID 27299675
- [Background] Kolka CM, Rattigan S, Richards SM, Barrett EJ, Clark MG. Endothelial Na+-D-glucose cotransporter: no role in insulin-mediated glucose uptake. Horm Metab Res. 2005 Nov;37(11):657-61. doi: 10.1055/s-2005-870574. PMID 16308832
- [Background] Chai W, Wang W, Liu J, Barrett EJ, Carey RM, Cao W, Liu Z. Angiotensin II type 1 and type 2 receptors regulate basal skeletal muscle microvascular volume and glucose use. Hypertension. 2010 Feb;55(2):523-30. doi: 10.1161/HYPERTENSIONAHA.109.145409. Epub 2009 Dec 7. PMID 19996061
- [Background] Wang N, Ko SH, Chai W, Li G, Barrett EJ, Tao L, Cao W, Liu Z. Resveratrol recruits rat muscle microvasculature via a nitric oxide-dependent mechanism that is blocked by TNFalpha. Am J Physiol Endocrinol Metab. 2011 Jan;300(1):E195-201. doi: 10.1152/ajpendo.00414.2010. Epub 2010 Oct 26. PMID 20978231
- [Background] Fu Z, Zhao L, Aylor KW, Carey RM, Barrett EJ, Liu Z. Angiotensin-(1-7) recruits muscle microvasculature and enhances insulin's metabolic action via mas receptor. Hypertension. 2014 Jun;63(6):1219-27. doi: 10.1161/HYPERTENSIONAHA.113.03025. Epub 2014 Apr 7. PMID 24711523
- [Background] Nalysnyk L, Hernandez-Medina M, Krishnarajah G. Glycaemic variability and complications in patients with diabetes mellitus: evidence from a systematic review of the literature. Diabetes Obes Metab. 2010 Apr;12(4):288-98. doi: 10.1111/j.1463-1326.2009.01160.x. PMID 20380649